CLINICAL TRIAL: NCT06648902
Title: A Phase 1/2 Study of the Safety and Preliminary Efficacy of Meldonium in Patients with Metastatic Renal Cell Carcinoma and Treatment-associated Fatigue.
Brief Title: Safety and Preliminary Efficacy of Meldonium in Patients with Metastatic Renal Cell Carcinoma and Treatment-associated Fatigue
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kidney Cancer Research Bureau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: KCRB-0102-MEL
Record Dates: First submitted 2024-09-22; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-09

CONDITIONS: Renal Cell Cancer Metastatic; Kidney Cancer; Fatigue Related to Cancer Treatment
MeSH Terms: conditions — Kidney Neoplasms | interventions — 3-(2,2,2-trimethylhydrazine)propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: First-line TKI therapy, Meldonium 500 mg (Experimental): meldonium 500 mg orally daily for six weeks.
  Interventions: Drug: meldonium
- Arm B: Second-line TKI therapy, Meldonium 1,000 mg (Experimental): meldonium 1,000 mg orally daily for six weeks.
  Interventions: Drug: meldonium
- Arm C: First-line IO-TKI therapy, Meldonium 1,000 mg (Experimental): meldonium 1,000 mg orally daily for six weeks.
  Interventions: Drug: meldonium

INTERVENTIONS:
Drug: meldonium — 500 mg (Arm A) or 1,000 mg (Arms B and C) orally daily, weeks 1-6

SUMMARY:
Fatigue is a prevalent adverse event associated with systemic therapy using tyrosine kinase inhibitors (TKIs). Meldonium, a fatty acid oxidation inhibitor, modifies the carnitine pathway, a nutrient critical for fat metabolism. The World Anti-Doping Agency (WADA) classified meldonium as a banned substance due to its documented use by athletes aiming to enhance physical performance. In this study, the safety and preliminary efficacy of meldonium in treatment-related fatigue will be assessed.

DETAILED DESCRIPTION:
Fatigue is a frequent symptom of cancer and the most common adverse event of treatment with tyrosine kinase inhibitors. For example, in phase 2 randomized study 59% of patients with metastatic renal cell carcinoma experienced any grade fatigue during treatment with the combination of lenvatinib and everolimus. Fourteen percent of patients had grade 3 fatigue or asthenia. Fatigue was also most frequently reported treatment-related adverse event in patients with unresectable hepatocellular carcinoma (30%), and advanced thyroid cancer (60%) treated with lenvatinib. Additionally, fatigue is one of the most common adverse events associated with the administration of checkpoint inhibitors. Frequency of fatigue was 55% in patients with endometrial cancer treated with combination of pembrolizumab and lenvatinib.

Meldonium is a fatty acid oxidation inhibitor, and it is now principally used for heart conditions, such as angina, heart attack, heart failure, and others. The compound works by altering pathways for carnitine, a nutrient involved in fat metabolism. Meldonium received the greatest fame in sport. The World Anti-Doping Agency (WADA) added meldonium to their list of banned substances in 2016 because of evidence of its use by athletes with the intention of enhancing performance. Center for Preventive Doping Research and European Monitoring Center for Emerging Doping Agents showed that mildronate demonstrates an increase in endurance performance of athletes, improved rehabilitation after exercise, protection against stress, and enhanced activations of the central nervous system functions. Based on these data, meldonium can be a possible option in cancer patients with fatigue treated with targeted or imminotargeted therapy. Moreover, the compound could decrease the number of vascular adverse events of TKIs.

ELIGIBILITY:
Inclusion Criteria:

* metastatic renal cell carcinoma
* measurable disease based on RECIST 1.1 criteria
* systemic therapy with targeted or immunotargeted therapy
* any grade of fatigue associated with targeted or immunotargeted therapy
* ECOG PS <2
* signed informed consent

Exclusion Criteria:

* Any treatment for fatigue
* Uncompensated hypothyroidism
* Anemia
* Pregnant or nursing
* Local and/or systemic infections requiring antibiotics or COVID-19 within 28 days prior to study entry
* Other malignancy
* Brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From enrollment to the end of treatment at 6 weeks
  Incidence of meldonium-related adverse events
Changes in fatigue levels based on FACIT Fatigue Scale | From enrollment to the end of treatment at 6 weeks
  Changes in fatigue levels, measured at six weeks using the FACIT Fatigue Scale (Version 4).

SECONDARY OUTCOMES:
Toxicity of anti-cancer systemic therapy | From enrollment to the end of treatment at 8 weeks
  Rate of adverse events
Rate of discontinuation of anti-cancer therapy and/or dose reduction of the drug | From enrollment to the end of treatment at 12 weeks
  Rate of discontinuation of anti-cancer therapy and/or dose reduction of the drug
Rate of arterial hypertension | From enrollment to the end of treatment at 12 weeks
  Rate of arterial hypertension as an adverse event of targeted therapy

CONTACTS AND LOCATIONS:
Locations (3):
- Megis medical clinic, Tirana, Albania
- National Center of Oncology, Baku, Azerbaijan
- STOONCO clinic, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided